CLINICAL TRIAL: NCT03762564
Title: A Randomized, Multicenter Open Label Phase II Trial of Paclitaxel + Ramucirumab Versus Paclitaxel Alone in Patients With Squamous-cell Carcinoma of the Esophagus, Refractory or Intolerant to Combination Therapy With Fluoropyrimidine and Platinum-based Drugs - The RAMOS STUDY
Brief Title: Study With Paclitaxel +/- Ramucirumab in Patients With Squamous-cell Carcinoma of the Esophagus After Prior Therapy
Acronym: RAMOS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest (Other)
Collaborators: Eli Lilly and Company (Industry); Trium Analysis Online GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RAMOS; AIO-STO-0216 (Other: AIO); 2016-003850-33 (EudraCT Number)
Record Dates: First submitted 2018-11-27; First posted 2018-12-03 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Squamous Cell Carcinoma of the Esophagus
Keywords: Squamous Cell Carcinoma of the Esophagus; Ramucirumab; Paclitaxel
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Ramucirumab; Paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Paclitaxel + Ramucirumab) (Experimental): Paclitaxel 80 mg/m2 as 1 hour intravenous infusion on day 1, 8, 15 plus Ramucirumab 8 mg/kg as 1 hour intravenous infusion on day 1 and 15 qd 28
  Interventions: Drug: Ramucirumab; Drug: Paclitaxel
- Arm B (control arm) (Active Comparator): Paclitaxel 80 mg/m2 as 1 hour intravenous infusion on day 1, 8, 15 qd 28
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Drug: Ramucirumab — Ramucirumab 8 mg/kg i.v. infusion on day 1 and 15
  Other Names: Cyramza
  Arms: Arm A (Paclitaxel + Ramucirumab)
Drug: Paclitaxel — Paclitaxel 80 mg/m2 on day 1, 8, 15

SUMMARY:
This is a multicenter, randomized, controlled, open-label phase II study including patients with squamous-cell carcinoma of the esophagus, refractory or intolerant to combination therapy with Fluoropyrimidine and Platinum-based drugs.

DETAILED DESCRIPTION:
This is a phase II, randomized, open-label multi-center study comparing treatment of paclitaxel plus ramucirumab with paclitaxel monotherapy in patients with advanced squamous-cell carcinoma (SCC) of the esophagus.

Adult patients with histologically or cytologically confirmed advanced squamous-cell carcinoma of the esophagus and refractory or intolerant to combination therapy with Fluoropyrimidine and Platinum-based drugs will be enrolled in the study.

A total number of 186 patients will be enrolled (Randomization 1:1). 93 patients will be treated with paclitaxel + ramucirumab (Arm A) and 93 with paclitaxel (Arm B).

Randomization will be stratified by time of progression during or after end of first-line therapy (≤3 months vs. >3 months).

The primary objective is to compare overall survival (OS) after 6 months in patients with squamous-cell carcinoma of the esophagus, refractory or intolerant to combination therapy with Fluoropyrimidine and Platinum-based drugs receiving paclitaxel with ramucirumab versus paclitaxel alone in the intent-to-treat population (ITT). OS is defined as the time from randomization to death from any cause.

Patients in Arm A (investigational arm) receive Paclitaxel 80 mg/m2 on day 1, 8, 15 plus Ramucirumab 8 mg/kg i.v. infusion on day 1 and 15 every 4 weeks. Patients in Arm B (control arm) receive Paclitaxel 80 mg/m2 on day 1, 8, 15 every 4 weeks. Study treatment will be continued until progression or intolerable toxicity, but for a maximum of 1 year.

Tumor assessment will be performed according to clinical routine at screening / baseline and every 8 weeks.

After discontinuation of study medication, patients will be followed for up to 1 year. Tumor assessments per CT or MRI will be performed every 2 months for 6 months or until documentation of disease progression. Follow-up for survival will be done and documented every 2 months for the 1 year follow-up period after end of treatment.

During treatment, clinical visits (blood cell counts, detection of toxicity) will be performed prior to every treatment dose. Safety of paclitaxel +/- ramucirumab will be monitored continuously by careful monitoring of all adverse events (AEs) and serious adverse events (SAEs) reported. Prior to the start of each cycle and at the 30-day safety follow-up visit Quality of life (QoL) will be assessed using the European Organization for Research and treatment of Cancer Quality of Life Questionnaire-C30 (EORTC-QLQ-C30).

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent;
2. Male or female* ≥ 18 years of age; Patients in reproductive age must be willing to use adequate contraception during the study and for 6 months after the end of ramucirumab treatment (Appropriate contraception is defined as surgical sterilization (e.g., bilateral tubal ligation, vasectomy), hormonal contraception (implantable, patch, oral), and double-barrier methods (any double combination of: IUD, male or female condom with spermicidal gel, diaphragm, sponge, cervical cap)). Female patients with childbearing potential need to have a negative pregnancy test within 7 days before study start.

   *There are no data that indicate special gender distribution. Therefore, patients will be enrolled in the study gender-independently.
3. Histologically proven squamous cell carcinoma of the esophagus

   * Adult patients with metastatic or locally advanced squamous-cell carcinoma of the esophagus, not amenable to potentially curative resection, who are refractory to or intolerant of prior platinum/fluoropyrimidine combination therapy. The definition of refractory should be defined as follows:
   * Patients whose PD or recurrence was confirmed by imaging during their initial chemotherapy (including chemoradiation) or within 8 weeks after the last dose of chemotherapy will be assessed as "refractory".
   * Patients after radical resection in conjunction with chemotherapy, including neoadjuvant/adjuvant therapy and chemoradiation, whose recurrence was confirmed by imaging within 24 weeks after the last dose of chemotherapy, will be determined "refractory".
4. Measurable or non-measurable but evaluable disease determined using guidelines in RECIST 1.1 as confirmed within 28 days before randomization
5. ECOG performance status 0-1;
6. Life expectancy > 12 weeks;
7. Adequate hematological, hepatic and renal functions:

   * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L;
   * Platelets ≥ 100 x 109/L;
   * Hemoglobin ≥9 g/dL (5.58 mmol/L
   * Total bilirubin ≤ 1.5 times the upper normal limit (UNL)
   * AST (SGOT) and ALT (SGPT) ≤ 2.5 x UNL in absence of liver metastases, or ≤ 5 x UNL in presence of liver metastases; AP ≤ 5 x UNL
   * Serum creatinine ≤ 1.5 x upper limit of normal, or creatinine clearance (measured via 24-hour urine collection) ≥40 mL/minute (that is, if serum creatinine is >1.5 times the ULN, a 24-hour urine collection to calculate creatinine clearance must be performed)
   * Urinary protein ≤1+ on dipstick or routine urinalysis (UA; if urine dipstick or routine analysis is ≥2+, a 24-hour urine collection for protein must demonstrate <1000 mg of protein in 24 hours to allow participation in this protocol).
   * Adequate coagulation function as defined by International Normalized Ratio (INR) ≤ 1.5, and a partial thromboplastin time (PTT) ≤ 5 seconds above the ULN (unless receiving anticoagulation therapy). Patients on full-dose anticoagulation must be on a stable dose (minimum duration 14 days) of oral anticoagulant or low molecular weight heparin (LMWH). Patients receiving warfarin/ phenprocoumon must be switched to low molecular weight heparin and have an INR ≤3.0 prior to first dose of protocol therapy. For heparin and LMWH there should be no active bleeding (that is, no bleeding within 14 days prior to first dose of protocol therapy) or pathological condition present that carries a high risk of bleeding (for example, tumor involving major vessels or known varices).
8. Ability to comply with scheduled assessments and with management of toxicities

Exclusion Criteria:

1. Other tumor type than squamous carcinoma (e.g. leiomyosarcoma, lymphoma) or a second cancer except in patients with squamous or basal cell carcinoma of the skin or carcinoma in situ of the cervix that has been effectively treated. Patients curatively treated and disease-free for at least 5 years will be discussed with the sponsor before inclusion.
2. Patients with significant malnutrition who receive intravenous hyperalimentation or require continuous infusion therapy with hospitalization.
3. Patients with apparent tumor invasion on organs located adjacent to the esophageal disease. Patients will be excluded if they are receiving stent therapy in esophagus or respiratory tract.
4. Concurrent chronic systemic immune therapy, chemotherapy, or hormone therapy not indicated in the study protocol.
5. Previous therapy with paclitaxeI
6. Current treatment with any anti-cancer therapy ≤ 2 weeks prior to study treatment start, unless rapidly progressing disease is measured
7. Concurrent treatment with any other anti-cancer therapy
8. Previous exposure to a VEGF or VEGFR inhibitor or any antiangiogenic agent, or prior enrolment in this study
9. Patient has undergone major surgery within 28 days prior to first dose of protocol therapy, or minor surgery/subcutaneous venous access device placement within 7 days prior to first dose of protocol therapy. The patient has elective or planned major surgery to be performed during the course of the clinical trial.
10. Grade 3-4 GI bleeding within 3 months prior to enrollment
11. History of deep vein thrombosis (DVT), pulmonary embolism (PE), or any other significant thromboembolism (venous port or catheter thrombosis or superficial venous thrombosis are not considered "significant") during the 3 months prior to first dose of protocol therapy-
12. Cirrhosis at a level of Child-Pugh B (or worse) or cirrhosis (any degree) and a history of hepatic encephalopathy or clinically meaningful ascites resulting from cirrhosis. Clinically meaningful ascites is defined as ascites from cirrhosis requiring diuretics or paracentesis.
13. Known brain or leptomeningeal metastases.
14. Known allergic/ hypersensitivity reaction to any of the components of the treatment.
15. Other serious illness or medical conditions within the last 12 months prior to study drug administration.
16. Any arterial thromboembolic events, including but not limited to myocardial infarction, transient ischemic attack, cerebrovascular accident, or unstable angina, within 6 months prior to first dose of protocol.
17. The patient has uncontrolled or poorly-controlled hypertension (>160 mmHg systolic or > 100 mmHg diastolic for >4 weeks) despite standard medical management.
18. Active uncontrolled infection.
19. Active disseminated intravascular coagulation.
20. Any other serious concomitant disease or medical condition that in the judgment of the investigator renders the subject at high risk of treatment complication or reduced the probability of assessing clinical effect
21. Prior history of GI perforation/fistula (within 6 months of first dose of protocol therapy) or risk factors for perforation.
22. Serious or nonhealing wound, ulcer, or bone fracture within 28 days prior to first dose of protocol therapy.
23. The patient is receiving chronic antiplatelet therapy, including aspirin, nonsteroidal anti-inflammatory drugs (NSAIDs, including ibuprofen, naproxen, and others), dipyridamole or clopidogrel, or similar agents. Once-daily aspirin use (maximum dose 325 mg/day) is permitted.
24. Concurrent treatment with other experimental drugs or participation in another clinical trial with any investigational drug within 30 days prior to treatment start.
25. Known drug abuse/ alcohol abuse.
26. Lack of resolution of all toxic effects (excluding alopecia) of prior chemotherapy, prior radiotherapy or surgical procedure to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) grade < 1. Note: Neuropathy due to prior chemotherapy is allowed if not > NCI Grade II according to CTCAE version 4.0.
27. Subject pregnant or breast feeding, or planning to become pregnant within 6 months after the end of treatment.
28. Subject (male or female) is not willing to use highly effective methods of contraception (per institutional standard) during treatment and for 6 months (male or female) after the end of treatment.
29. Patients with a psychiatric illness or patients imprisoned or working in the institution of the treating physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-03-08 (Actual); Primary Completion 2022-07-04 (Actual); Study Completion 2022-11-25 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) at 6 months | 6 months
  OS rate at 6 months, defined as patients who are alive after at 6 months

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to 2 years
  PFS, defined as the time from randomization to the first occurrence of progression, as determined by the investigator using CT criteria, or death from any cause
Overall survival | Up to 2 years
  Overall survival according to Kaplan-Meier
Objective response rate | Up to 2 years
  Objective response rate defined as the proportion of patients with complete or partial remission according to RECIST 1.1
Tumor control rate | Up to 2 years
  Tumor control rate defined as the proportion of patients with complete or partial remission or stable disease according to RECIST 1.1
Quality of life (QoL) | Up to 1 year and 30 days
  Quality of life (QoL) as measured by EORTC-QLQ-C30 at d1 of each cycle, on EOT (end of treatment) and 30 days after EOT.
Incidence and severity of adverse events | Up to 1 year and 30 days
  incidence and severity of adverse events according to CTCAE (Common Terminology Criteria for Adverse Events) Version 4 criteria as assessed at day 1, 8 and 15 of every cycle during treatment for a maximum of 12 months and until 30 days after the last dose of study drug

CONTACTS AND LOCATIONS:
Overall Officials: Salah-Eddin Al-Batran, Prof. Dr., Study Chair — Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest
Locations (2):
- Germany (2):
  - Institute for Clinical Cancer Research Krankenhaus Nordwest, Frankfurt
  - Technische Universität München Klinikum rechts der Isar, München

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared